CLINICAL TRIAL: NCT06959290
Title: Effect of Multiple Non-pharmacological Methods for Pain Management During Eye Examination for Retinopathy of Prematurity in Preterm Infants: A Randomised Controlled Crossover Trial
Brief Title: Effect of Multiple Non-pharmacological Methods for Pain Management During Eye Examination for Retinopathy of Prematurity in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Aynur Aytekin Ozdemir, Professor, Istanbul Medeniyet University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 01.11.2024/21
Record Dates: First submitted 2025-04-28; First posted 2025-05-06 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Premature Infant; Retinopaty of Prematurity; Pain Management
Keywords: Premature Infant; Retinopaty of prematurity examination; Pain management
MeSH Terms: conditions — Premature Birth; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Sham Comparator): Retinopathy of prematurity examination will be performed according to clinical routine practice.
  Interventions: Other: Routine Treatment
- Intervention Group (Active Comparator): Multiple nonpharmacological methods will be applied for pain management during retinopathy of prematurity examination.
  Interventions: Procedure: Multiple nonpharmacological methods

INTERVENTIONS:
Procedure: Multiple nonpharmacological methods — The preterm babies in this group are swaddled by the nurse with each baby's own blanket 2 minutes before the ROP examination. The nurse will then give the baby 25% dextrose solution orally (0.5ml for those <32 weeks gestation, 1ml for those >32 weeks gestation). The nurse then places a pacifier soaked in 25% dextrose solution in the preterm infant's mouth. After these three non-pharmacological methods, the doctor will perform the ROP examination.
  Arms: Intervention Group
Other: Routine Treatment — The preterm babies in this group are swaddled by the nurse with each baby's own blanket 2 minutes before the ROP examination. After these three non-pharmacological methods, the doctor will perform the ROP examination.
  Arms: Control Group

SUMMARY:
This study will be conducted to determine the effect on pain and vital signs of multiple nonpharmacological methods used in preterm infants during the examination for retinopathy of prematurity (ROP).

DETAILED DESCRIPTION:
Retinopathy of prematurity (ROP) examination is performed using a binocular indirect ophthalmoscope. ROP examination causes pain and discomfort in the preterm infant in many ways, including the application of eye drops, the placement of the speculum in the eye, the pressure applied to the pupils and the brightness of the ophthalmoscope. Studies in the literature have also reported that newborns experience pain and discomfort during ROP examination. In relation to the ROP pain experienced by the preterm infant, various physiological changes such as increased heart rate or decreased oxygen saturation are experienced during or after the examination. Accordingly, ROP examination is important; however, controlling the pain that occurs during the examination is also very important in terms of the patient's emotional experience and comfort. In the literature, many studies have been conducted to reduce pain during ROP examination. Although pharmacological treatment methods are an effective technique to reduce pain, it is recommended that nonpharmacological methods should be used especially in infants and children because of the side effects of drugs (such as apnoea, bradycardia, respiratory depression, hypotension) and the method to be used should be easy, fast and does not require preparation. The Turkish Neonatology Society and the Turkish Ophthalmology Society also recommend that ROP examination is a very painful procedure, that pharmacological methods alone are not sufficient to reduce pain, and that nonpharmacological methods such as pacifier, breast milk and oral sucrose should be used during the examination. In addition, although there is no gold standard for pain relief during ROP examination, previous studies suggest that clinicians should use more than one method together to reduce pain and provide relief in premature infants. In this study, a combination of oral 25% dextrose, non-nutritive sucking and swaddling will be used for multiple nonpharmacological applications

ELIGIBILITY:
Inclusion Criteria:

* Postmenstrual gestational age ≤32 weeks and/or birth weight ≤1500 g,
* Stable, awake, in supine position and breathing spontaneously without oxygen support,
* Vital signs were within normal limits before the examination,
* Premature infants undergoing ROP examination for the first time.

Exclusion Criteria:

* Preterms who have been administered non-steroidal anti-inflammatory drugs or sedative and antiepileptic drugs such as chloral hydrate, phenobarbital and diazepam within 24 hours before the ROP examination,
* Preterms with severe respiratory diseases, receiving respiratory support (continuous positive airway pressure or mechanical ventilation),
* Preterms with critical conditions such as central nervous system infections and sepsis,
* Preterms with other organic diseases such as severe cardiovascular disease, pulmonary insufficiency,
* Preterms with congenital malformations.

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Procedural pain score: Premature Infant Pain Profile-Revised Scale (PIPP-R) | 1 minute before the procedure, during the procedure, 2 minutes after the procedure and 5 minutes after the procedure
  The PIPP-R is a seven indicator composite pain measure consisting of three behavioural (facials actions of brow bulge, eye squeeze, naso-labial furrow), two physiological (heart rate, oxygen saturation), and two contextual (gestational age, behavioural state) indicators validated for pain measurement in infants 26-44 weeks' gestation. A score of <7 is indicative of minimal pain and a score ≥ 12 is indicative of moderate to severe pain.

SECONDARY OUTCOMES:
Oxygen saturation | 1 minute before the procedure, during the procedure, 2 minutes after the procedure and 5 minutes after the procedure
  Premature infants will be connected to a pulse oximeter monitor; oxygen saturation will be monitored before, during and after the procedure.
Heart rate | 1 minute before the procedure, iduring the procedure, 2 minutes after the procedure and 5 minutes after the procedure
  Premature infants will be connected to a pulse oximeter monitor; heart rate will be monitored before, during and after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Aynur Aytekin Ozdemir, Professor, Study Director — İstanbul Medeniyet University
Locations (1):
- Istanbul Medeniyet University, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.
Supporting Information: Study Protocol
Time Frame: July through December of 2026
Access Criteria: Individual participant data may be shared upon request from the principal investigator, subject to the appropriateness of the request, while ensuring adherence to the rules of confidentiality regarding individual data.